CLINICAL TRIAL: NCT03030599
Title: A Double-Blind, Placebo-Controlled, Randomized-Withdrawal, Multicenter Study of the Efficacy and Safety of JZP-258 in Subjects With Narcolepsy With Cataplexy
Brief Title: A Study of the Efficacy and Safety of JZP-258 in Subjects With Narcolepsy With Cataplexy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-006; 2016-000426-20 (EudraCT Number)
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Narcolepsy With Cataplexy
MeSH Terms: conditions — Narcolepsy | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- JZP-258 (Experimental): JZP-258
  Interventions: Drug: JZP-258

INTERVENTIONS:
Drug: JZP-258 — JZP-258 oral solution 0.5 g/mL, which is equivalent to 0.413 g/mL of oxybate
  Other Names: Xyrem®
  Arms: JZP-258
Other: Placebo — Matching placebo solution (aqueous solution containing sodium citrate, malic acid, and sucralose; all ingredients were compendial [United States Pharmacopeia/ National Formulary])
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomized-withdrawal, multicenter study of the efficacy and safety of JZP-258.

DETAILED DESCRIPTION:
Subjects will be transitioned to JZP-258 based on their treatment status at study entry. All subjects will begin JZP-258 treatment at the beginning of this period and continue through Week 12. They will be treated with JZP-258 alone for the final two weeks of this 12-week period. Once the JZP-258 dose has been optimized per the Investigator's judgment, these subjects may enter the 2-week Stable-Dose Period with that dose. Subjects are eligible to enter the Double-Blind Randomized-Withdrawal Period if the dose of JZP-258 remains unchanged during the Stable-Dose Period and, in the judgment of the Investigator, no clinically significant worsening in narcolepsy symptoms or clinically significant adverse events due to JZP-258 treatment have occurred. Subjects will return for a Safety Follow-up visit 2 weeks after the Double-Blind Randomized-Withdrawal Period. Subjects who complete the double-blind treatment period during the Main Study are eligible to enter a 24-week Open-Label Extension. During this period subjects will receive open label JZP-258. Subjects will return for a Safety Follow-up visit 2 weeks after the Open-Label Extension Period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 70 years of age, inclusive.
2. Have a primary diagnosis of narcolepsy with cataplexy that meets ICSD-3 criteria or DSM-5 criteria, and currently untreated or treated with or without anticataplectics.
3. If applicable, treated with a stimulant or alerting agent at unchanged doses for at least 2 months prior to dosing or not treated with a stimulant or alerting agent.
4. Willing and able to comply with the study design schedule and other requirements.
5. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Narcolepsy secondary to another medical condition (e.g., CNS injury or lesion)
2. History or presence of any unstable or clinically significant medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or history or presence of another neurological disorder or surgical history that might affect the subject's safety and/or interfere with the conduct of the study in the opinion of the Investigator.
3. Treatment with any central nervous system sedating agents, including but not limited to benzodiazepines, nonbenzodiazepine anxiolytics/ hypnotics/sedatives, neuroleptics, opioids, barbiturates, phenytoin, ethosuximide, or MCT inhibitors, e.g. diclofenac, valproate, ibuprofen, within 2 weeks prior to enrollment (discontinuation for the purpose of study enrollment is permitted only if considered safe by the Investigator and approved by the Medical Monitor).
4. Treatment with an antidepressant for cataplexy, if the withdrawal of the antidepressant during cross-titration with JZP-258 might be unsafe due to prior history of depression.
5. Unsafe for the subject to receive placebo treatment for 2 weeks, in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trial Disclosure & Transparency, Study Director — Jazz Pharmaceuticals
Locations (25):
- United States (12):
  - SDS Clinical Trials, Inc., Orange, California
  - Stanford Health Services, Stanford, California
  - Colorado Sleep Institute, Boulder, Colorado
  - Pulmonary Disease Specialists, Kissimmee, Florida
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Kentucky Research Group, Louisville, Kentucky
  - Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Montefiore/ Sleep-Wake Disorders Center, The Bronx, New York
  - Gastonia Medical Specialty Clinic, Gastonia, North Carolina
  - Research Carolina, Huntersville, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - Cleveland Clinic, Sleep Disorder Center, Cleveland, Ohio
- Belgium (3):
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Czechia (2):
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
- Helsingin Uniklinikka, Vitalmed Oy, Helsinki, Finland
- France (2):
  - Hôpital Gui de Chauliac, Montpellier, Herault
  - Hopital Roger Salengro - CHU Lille, Lille
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General de Castellón, Castelló
  - Instituto de Investigaciones del Sueño, Madrid
  - Hospital Vithas Nuestra Señora de America, Madrid

REFERENCES:
- [Derived] Bogan RK, Foldvary-Schaefer N, Skowronski R, Chen A, Thorpy MJ. Long-Term Safety and Tolerability During a Clinical Trial and Open-Label Extension of Low-Sodium Oxybate in Participants with Narcolepsy with Cataplexy. CNS Drugs. 2023 Apr;37(4):323-335. doi: 10.1007/s40263-023-00992-y. Epub 2023 Mar 22. PMID 36947322
- [Derived] Dauvilliers Y, Sonka K, Bogan RK, Partinen M, Del Rio Villegas R, Foldvary-Schaefer N, Skowronski R, Chen A, Black J, Skobieranda F, Thorpy MJ. Changes in Cataplexy Frequency in a Clinical Trial of Lower-Sodium Oxybate with Taper and Discontinuation of Other Anticataplectic Medications. CNS Drugs. 2022 Jun;36(6):633-647. doi: 10.1007/s40263-022-00926-0. Epub 2022 May 30. PMID 35635687
- [Derived] Bogan RK, Thorpy MJ, Dauvilliers Y, Partinen M, Del Rio Villegas R, Foldvary-Schaefer N, Skowronski R, Tang L, Skobieranda F, Sonka K. Efficacy and safety of calcium, magnesium, potassium, and sodium oxybates (lower-sodium oxybate [LXB]; JZP-258) in a placebo-controlled, double-blind, randomized withdrawal study in adults with narcolepsy with cataplexy. Sleep. 2021 Mar 12;44(3):zsaa206. doi: 10.1093/sleep/zsaa206. PMID 33184650

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were evaluated for eligibility during the Screening Period (up to 30 days).
Groups:
- Open-label JZP-258: All 201 subjects entered the Open Label Optimized Treatment and Titration Period (OL OTTP) and received at least 1 dose of study drug. During the OL OTTP (12 weeks), eligible subjects were transitioned to JZP-258 treatment based on their pre-treatment status. During the Stable Dose Period, subjects received open-label JZP-258 at the same unchanged dose that they received during the last 2 weeks of the Open Label Treatment and Titration Period.
- JZP-258: JZP-258 at the dose taken during the last 2 weeks of the Stable Dose Period.
- Placebo: A matching oral solution to JZP-258.
Period: Open Label Treatment and Titration
Arm/Group | Open-label JZP-258 | JZP-258 | Placebo
Started | 201 | 0 | 0
Completed | 155 | 0 | 0
Not Completed | 46 | 0 | 0
Not completed — Protocol deviation | 8 | 0 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Non-Compliance with Study Drug | 4 | 0 | 0
Not completed — Adverse Event | 18 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Sponsor decision | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Period: Stable Dose
Arm/Group | Open-label JZP-258 | JZP-258 | Placebo
Started | 149 (149 subjects of the 201 entered the Stable Dose Period. Of those subjects, 136 were randomized.) | 0 | 0
Completed | 144 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Protocol deviation | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Double Blind Randomized Withdrawal
Arm/Group | Open-label JZP-258 | JZP-258 | Placebo
Started | 0 | 69 (134 of the 136 subjects randomized received at least 1 dose of study drug in the DB RWP.) | 67 (134 of the 136 subjects randomized received at least 1 dose of study drug in the DB RWP.)
Completed | 0 | 69 | 59
Not Completed | 0 | 0 | 8
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Randomized in error | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Open-label Extension
Arm/Group | Open-label JZP-258 | JZP-258 | Placebo
Started | 74 | 0 | 0
Completed | 67 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Other Reason | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label Treatment and Titration: All 201 subjects entered the Open Label Optimized Treatment and Titration Period (OL OTTP) and received at least 1 dose of study drug. During the OL OTTP (12 weeks), eligible subjects were transitioned to JZP-258 treatment based on their pre-treatment status. During the Stable Dose Period, subjects received open-label JZP-258 at the same unchanged dose that they received during the last 2 weeks of the Open Label Treatment and Titration Period.
Arm/Group | Open Label Treatment and Titration
Number analyzed (Participants) | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 195
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 177
  More than one race | 2
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Number of Cataplexy Attacks
Description: Participants completed a daily Cataplexy Frequency Diary each night prior to bedtime. Participants were to record the number of cataplexy attacks that they had each day.
Time Frame: Change from baseline (2 weeks of the Stable Dose Period) to the 2 weeks of the Double Blind Randomized Withdrawal Period (DB RWP)
Population: The efficacy population contains all randomized subjects who received at least one dose of double-blind study drug and had at least one set of post-randomization efficacy data.
Measure: Median (Inter-Quartile Range); unit: attacks
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 69 | 65
attacks | 0.00 [-0.49 to 1.75] | 2.35 [0.00 to 11.61]

2. Secondary Outcome: Change in the Epworth Sleepiness Scale (ESS) Score
Description: This is the key secondary endpoint. The Epworth Sleepiness Scale (ESS) was a self-administered questionnaire with 8 questions. Participants were asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most participants engaged in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that participants average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Time Frame: From the end of the Stable Dose Period to the end of the Double Blind Randomized Withdrawal Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 69 | 65
score on a scale | 0.00 [-1.0 to 1.0] | 2.0 [0.00 to 5.0]

3. Secondary Outcome: Number of Participants With Worsening Patient Global Impression of Change (PGIc) for Narcolepsy Overall
Description: At the end of the Double Blind Randomized Withdrawal Period (DB RWP), participants rated the change in their condition on a 7-point scale ranging from 1 = "very much improved" to 7 = "very much worse" since the last visit. This endpoint measures the percentage of participants with worsening PGIc scores for narcolepsy overall (defined as scores of Much Worse or Very Much Worse).
Time Frame: At the end of the Double Blind Randomized Withdrawal Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 69 | 65
Participants | 3 | 29

4. Secondary Outcome: Number of Participants With Worsening Clinical Global Impression of Change (CGIc) for Narcolepsy Overall
Description: At the end of the Double Blind Randomized Withdrawal Period, Investigators rated their impression of any change in the severity of the participant's narcolepsy overall condition since the start of the Double Blind Randomized Withdrawal Period on a 7-point scale ranging from 1 = "very much improved" to 7 = "very much worse". This endpoint measures the percentage of participants with worsening CGIc scores for narcolepsy overall, defined as scores of Much Worse or Very Much Worse.
Time Frame: At the end of the Double Blind Randomized Withdrawal Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 68 | 65
Participants | 4 | 39

5. Secondary Outcome: Change in 36-Item Short Form Health Survey Version 2 (SF-36v2) Scores
Description: The SF-36v2 is a multi-purpose, short-form health survey with 36 questions/ items. It yields an 8-scale profile of functional health and well-being scores as well as a psychometrically-based physical and mental overall component summary measures. Two summary scores were derived using the SF-36v2. Physical Component Summary measures dimensions of functional health that are meaningful to respondents, including the impact of health and health-related changes on physical function, pain, and the ability to carry out daily roles. The Mental Component Summary component scale measures the impact of health and health-related changes on well-being, including vitality, social function, and emotional well-being. Participants self-report on items in a summary that have between 2-6 choices per item (e.g. none of the time, some of the time, etc.). Summations of item scores were transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. Higher scores indicate better health status.
Time Frame: At the End of the Stable Dose Period to the End of the Double Blind Randomized Withdrawal Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 67 | 65
score on a scale
  Physical Component Summary | -0.03 [-2.07 to 2.41] | -1.92 [-3.46 to 1.73]
  Mental Component Summary | 1.55 [-1.88 to 3.78] | -1.92 [-6.28 to 1.34]

6. Secondary Outcome: Change in 5-level EQ-5D (EQ-5D-5L) Crosswalk Index Score and Visual Analog Scale
Description: The EQ-5D-5L is a measure of health outcome that includes a descriptive system consisting of 5 dimensions (mobility, self-care, usual activities, pain/ discomfort, and anxiety/ depression). The EQ-5D-5L includes 5 levels of severity for each of the 5 dimensions of the descriptive system (1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems) that reflect increasing levels of difficulty. The 5 digit health states for each dimension are converted into a single value per country (0= equivalent to death, 1= equivalent to best imaginable health and values below 0= health states rated worse than death capped at -1), using the EQ-5D-5L crosswalk index value calculator as recommended by EuroQol group. A visual analogue scale (VAS) used within this scale recorded the participants self-rated health on a VAS and the endpoints resulted in a numeric value set ranging from 0 (= worst imaginable health state) up to 100 (= best imaginable health state).
Time Frame: At the End of the Stable Dose Period to the End of the Double Blind Randomized Withdrawal Period
Population: There were 68 JZP-258 participants included in the Crosswalk Index, and 69 JZP-258 participants in the VAS Score. The efficacy population contains all randomized subjects who received at least one dose of double-blind study drug and had at least one set of post-randomization efficacy data.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | JZP-258 | Placebo
Number analyzed (Participants) | 69 | 65
score on a scale
  Crosswalk index: number analyzed (Participants) | 68 | 65
  Crosswalk index | 0.00 [-0.01 to 0.03] | 0.00 [-0.05 to 0.03]
  VAS Score | 0.00 [0.00 to 5.00] | -5.00 [-10.00 to 5.00]

ADVERSE EVENTS:
Time Frame: Through week 18 or early termination.
Description: Safety data are summarized for all subjects who received at least 1 dose of study medication across all periods.
Arm/Group | JZP-258 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/65
Serious Adverse Events (participants affected / at risk) | 5/201 | 2/65
Other Adverse Events (participants affected / at risk) | 108/201 | 12/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-258 (N=201) | Placebo (N=65)
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Muscle enzyme increased (Investigations) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral nerve paresis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Viral cardiomyopathy (Infections and infestations) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-258 (N=201) | Placebo (N=65)
Cataplexy (Nervous system disorders) | 21 | 5
Dizziness (Nervous system disorders) | 23 | 0
Headache (Nervous system disorders) | 45 | 1
Somnolence (Nervous system disorders) | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 27 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 1
Influenza (Infections and infestations) | 17 | 1
Nasopharyngitis (Infections and infestations) | 19 | 2
Upper respiratory tract infection (Infections and infestations) | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03030599/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03030599/SAP_003.pdf